CLINICAL TRIAL: NCT02767063
Title: Candidate Therapies in Combination or Sequentially With Tyrosine Kinase Inhibitors in Chronic Phase-chronic Myelogenous Leukemia Patients in CCR Without Achieving a Deep Molecular Response: an Adaptative Trial Based on a Drop Loser Design
Brief Title: Therapies in Combination or Sequentially With Tyrosine Kinase Inhibitors (TKIs) in Chronic Phase Chronic Myelogenous Leukemia Patients in CCR (ACTIW)
Acronym: ACTIW
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Clinical coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P13/12_ACTIW
Record Dates: First submitted 2016-03-16; First posted 2016-05-10 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Pioglitazone; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental Arm_ACTOS (Experimental): TKI : Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months
  PIOGLITAZONE (Actos®):
  30 mg per day for 12 months. The dose will be increased to 45 mg per day after 2 months in the absence of grade >1 related AE.
  Interventions: Drug: Pioglitazone
- controled Arm (No Intervention): TKI : Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months
- Experimental Arm_AVELUMAB (Experimental): TKI : Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months AVELUMAB: 10mg/kg every 2 weeks, for a maximum of 8 IV infusions over a 4 months' period.(If MR4.5 is acheived by the first 3 months the 7th and 8th infusions will be omitted)
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Pioglitazone — PIOGLITAZONE (Actos®): 30 mg per day for 12 months. The dose will be increased to 45 mg per day after 2 months in the absence of grade >1 related AE.
  Arms: Experimental Arm_ACTOS
Drug: Avelumab — 10mg/kg every 2 weeks, for a maximum of 8 IV infusions over a 4 months' period. (If MR4.5 is acheived by the first 3 months the 7th and 8th infusions will be omitted)
  Arms: Experimental Arm_AVELUMAB

SUMMARY:
Patients will be randomized in phase II trials to continue on the same TKI versus one of the alternative treatment approaches. If a patient is not eligible for one of the treatments, he (she) will be randomized between the options for which he (she) is eligible.

The trial will start with current available treatment options (experimental arms). New available treatment options may be open at any times later on. Authorized TKIs are imatinib, nilotinib, dasatinib, bosutinib and ponatinib.

For all options the treatment duration is for a minimum of 12 months and will be continued in the absence of adverse events following investigator decision. Each therapeutic option will be detailed in term of combination modalities, dose, dose adaptation, specific warnings, specific exclusion and inclusion criteria. The decision to introduce a new option will depend on the general pace of recruitment and on the assessment of the potential efficacy and safety of the new treatment, and will be implemented after scientific review by a protocol amendment.

Primary objective:

A. To select molecules in combination or sequentially with imatinib, nilotinib, dasatinib, bosutinib or ponatinib potentially able to produce a 25% increase in the Cumulative Incidence of MR4.5 as compare to control.

Secondary objectives:

A. To determine the safety of selected therapies

B. To determine the rate of MR4 by 12, 24, 36, 48 months in experimental and control arms

C. To determine the rates of MR4.5 by 24, 36, 48 months in experimental and control arms

D. To determine the rate of undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 12, 24, 36, 48 months in experimental and control arms

E. To estimate treatment free remission (TFR) in patients eligible for discontinuation studies

F. To investigate the relationship between biological activity and the clinical efficacy of the selected therapies

G. To assess the effects of the treatments on the number and clonogenicity of CML stem cells and other biological markers of interest

H. To estimate duration of response, progression-free survival, event free survival and overall survival.

DETAILED DESCRIPTION:
Patients will be randomised to continue on TKI (same daily dose) versus one of the alternative novel treatment approaches. If a patient is not eligible for one of the treatments, he can be randomised for the options for which he is eligible. All treatment options may be open at all times. Investigators must specify before randomization for which treatment option they want their patient be included and randomized.

Perspectives New treatment options will be introduced over time. The decision to introduce a new option will depend on the general pace of recruitment and the assessment of the potential efficacy and safety of the new treatment in this patient population, and will be implemented after scientific review by a protocol amendment.

The available treatment arms are:

1. TKI alone same daily dose (control arm)
2. TKI in combination with pioglitazone
3. TKI in combination with Avelumab (anti-PD-L1 antibody)

Planned treatment arms for the future may be :

1. TKI in combination with pegylated interferon
2. TKI in combination with arsenic trioxide
3. TKI in combination with Homoharringtonine

Protocol plan:

1. Control arm (Imatinib, nilotinib, dasatinib, bosutinib or ponatinib):

   Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months
2. Pioglitazone arm

   * TKI : Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months
   * PIOGLITAZONE (Actos®):

     30 mg per day for 12 months. The dose will be increased to 45 mg per day after 2 months in the absence of grade >1 related AE.
   * After 12 Months :

   Continue TKI at the same daily dose and STOP pioglitazone.
3. AVELUMAB arm

   * TKI : Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months
   * AVELUMAB: 10mg/kg every 2 weeks, for a maximum of 8 IV infusions over a 4 months' period. (If MR4.5 is acheived by the first 3 months the 7th and 8th infusions will be omitted)
   * After 12 Months :Continue TKI at the same daily dose.
4. Other experimental arm TKI : Daily dose and schedule identical to the daily dose and schedule administered during the last 3 months

   * Arsenic trioxide : to be determined after amendment
   * Pegylated Interferon : to be determined after amendment
   * Homoharringtonine : to be determined after amendment
   * Drug X
   * Drug Y

ELIGIBILITY:
Common Inclusion Criteria:

1. Patient aged 18y or more
2. Signed informed consent
3. Patient with Philadelphia chromosome positive chronic phase CML and M BCR-ABL1 transcript positivity at diagnosis
4. Treatment with imatinib, nilotinib, dasatinib or bosutinib for more than 2 years overall
5. No switch between tyrosine kinase inhibitors within the last 3 months
6. No dose modification within the last 3 months
7. Complete cytogenetic response or BCR-ABL1IS ≤ 1%
8. Detectable BCR-ABL1 with BCR-ABL1IS > 0.0032% (less than MR4.5)
9. ECOG grade 0 to 2
10. ASAT and ALAT ≤ 2.5 N
11. Bilirubin in serum ≤ 2.5 N
12. Men and Women of childbearing potential must be using an adequate method of contraception

These specific inclusion criteria will apply for the Avelumab arm in addition to the common criteria.

1. Hematologic:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L,
   2. Platelet count ≥ 100 × 109/L,
   3. Hemoglobin ≥ 9 g/dL. (may have been transfused).
2. Hepatic:

   a. Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range.
3. Renal: Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
4. Pregnancy test: Negative serum or urine pregnancy test at screening for women of childbearing potential.
5. Contraception: Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last Avelumab treatment administration if the risk of conception exists.

Common Exclusion Criteria:

1. Pregnant or lactating women,
2. Participation in another clinical trial with any investigative drug within 30 days prior to study enrolment,
3. Prior history of hematopoietic stem cell transplantation (autologous or allogenic)
4. Cardiovascular disease:

   * Stage II to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA) classification system for heart failure.
   * Myocardial infarction within the previous 6 months
   * Symptomatic cardiac arrhythmia requiring treatment
5. Grade III or IV fluid retention
6. Known BCR-ABL kinase domain mutation
7. CML patient not in chronic phase at diagnosis
8. Individuals with an active malignancy
9. Known HIV-positivity

These specific exclusion criteria will apply for the pioglitazone arm in addition to the common criteria.

1. Known osteoporosis with curative therapy (prophylactic therapy is not an exclusion criteria)
2. Patient requiring anti-diabetic medication

These specific exclusion criteria will apply for the Avelumab arm in addition to the common criteria:

1. IMMUNOSUPRESSANTS: Current use of immunosuppressive medication, EXCEPT for the following:

   1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
   2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
2. AUTOIMMUNE DISEASE: Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
3. ORGAN TRANSPLANTATION: Prior organ transplantation including allogenic stem-cell transplantation.
4. INFECTIONS: Active infection requiring systemic therapy.
5. HIV/AIDS: Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
6. HEPATITIS: Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
7. VACCINATION: Vaccination within 4 weeks of the first dose of Avelumab and while on trials is prohibited except for administration of inactivated vaccines
8. HYPERSENSITIIVTY TO STUDY DRUG: Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions tomonoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
9. CARDIOVASCULAR DISEASE: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia equiring medication.
10. OTHER PERSISTING TOXICITIES: Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
11. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of patients achieving a deep molecular response | 12 months
  The cumulative incidence of patients achieving a deep molecular response defined by MR4.5 or deeper (BCR-ABLIS ≤ 0.0032 %) by 12 months

SECONDARY OUTCOMES:
Adverse events | 12 Months
  Adverse events
The cumulative rate of patients achieving MR4.5 by 24months in experimental and control arms | 24 months
  The cumulative rate of patients achieving MR4.5 by 24months in experimental and control arms
The cumulative rate of patients achieving MR4.5 by 36 months in experimental and control arms | 36 months
  The cumulative rate of patients achieving MR4.5 by 36 months in experimental and control arms
The cumulative rate of patients achieving MR4.5 by 48 months in experimental and control arms | 48 months
  The cumulative rate of patients achieving MR4.5 by 48months in experimental and control arms
The cumulative rate of patients achieving MR4 by 12months in experimental and control arms | 12 months
  The cumulative rate of patients achieving MR4 by 12,months in experimental and control arms
The cumulative rate of patients achieving MR4 by 24 months in experimental and control arms | 24 months
  The cumulative rate of patients achieving MR4 by 24 months in experimental and control arms
The cumulative rate of patients achieving MR4 by 36 months in experimental and control arms | 36 months
  The cumulative rate of patients achieving MR4 by 36 months in experimental and control arms
The cumulative rate of patients achieving MR4 by 48 months in experimental and control arms | 48 months
  The cumulative rate of patients achieving MR4 by 48 months in experimental and control arms
The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 12months in experimental and control arms | 12 months
  The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 12months in experimental and control arms
The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 24months in experimental and control arms | 24 months
  The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 24, months in experimental and control arms
The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 36 months in experimental and control arms | 36 months
  The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 36 months in experimental and control arms
The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 48 months in experimental and control arms | 48 months
  The cumulative rate of patients with undetectable BCR-ABL1 transcript (sensitivity 40000 ABL copies) by 48 months in experimental and control arms
The rate of patients in treatment free remission during follow-up | 48 months
  The rate of patients in treatment free remission during follow-up
Quantification of CML- and normal-CFU in bone marrow by clonogenic assays and RTQ- PCR | 12 months
Survival | 48 months
  Survival
duration of response | 48 months
  duration of response
event free survival | 48 months
  event free survival
progression free survival | 48 months
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROUSSELOT, Principal Investigator — CH Versailles
Locations (23):
- France (23):
  - Martine GARDEMBAS, Angers
  - Pascale CONY.MAKHOUL, Annecy
  - Thorsten BRAUN, Bobigny
  - Etienne, Bordeaux
  - CHU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - CH Henri Mondor, Créteil
  - Rousselot, Le Chesnay
  - CHU Lille, Lille
  - CHU de LIMOGES, Limoges
  - Franck NICOLINI, Lyon
  - Institut P Calmette, Marseille
  - Viviane DUBRUILLE, Nantes
  - Hopital l'Archet, Nice
  - Eric JOURDAN, Nîmes
  - Hôpital La Source, Orléans
  - Delphine REA _St louis, Paris
  - Simona LAPUSAN_St Antoine, Paris
  - Cayssials, Poitiers
  - CHU de Rennes - Pontchaillou, Rennes
  - Hôpital René Huguenin, Saint-Cloud
  - Institut Universitaire contre le Cancer, Toulouse
  - CHU Tours, Tours